CLINICAL TRIAL: NCT06827522
Title: Analysis of the Effect of Skin-to-skin Contact with the Mother on Galvanic Skin Response Signals in Newborns
Brief Title: The Effect of Skin-to-skin Contact Between Mother and Newborn
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Fatma Ozdemir, Principal Investigator, Medical Doctor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024/224
Record Dates: First submitted 2025-02-04; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Galvanic Skin Response; Skin to Skin Contact
Keywords: Spinal anesthesia; General anesthesia; Skin to skin contact; Newborn

STUDY DESIGN:
Intervention Model Description: In the study, 100 volunteers (n=50 general anesthesia, n=50 spinal anaesthesia) will undergo caesarean section, and the choice of anaesthesia will be made with the consent of the patient. The type of anesthesia will evaluate the effects of skin-to-skin contact on the mother and baby..
  Prenatal GSR electrodes will be connected and signal recordings will be obtained from mother and baby, and the physiological effects of skin-to-skin contact will be analysed. APGAR score (Activity, pulse, grimace, apperarance, respiration 0-10), cord pH, birth weight and neonatal follow-up data will be recorded.
  GSR signals will be recorded and filtered with BIOPAC, features will be extracted and time and frequency analyses will be performed. Classification will be performed with artificial neural networks and deep learning.
  The results will be evaluated with statistical tests and the effect of anaesthesia type and skin-to-skin contact on mother-infant will be investigated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- General Anesthesia (Experimental): Pregnant women who will have a cesarean section under general anesthesia.
  Interventions: Procedure: Birth Under General Anesthesia
- Spinal Anestesia (Experimental): Pregnant women who will have a cesarean section under spinal anesthesia.
  Interventions: Procedure: Birth Under Spinal Anesthesia

INTERVENTIONS:
Procedure: Birth Under General Anesthesia — Before anaesthesia, GSR electrodes will be connected and signal recording will be started. After caesarean section, the newborn will be evaluated and GSR signals will be recorded again after the mother wakes up by providing skin-to-skin contact.
  Arms: General Anesthesia
Procedure: Birth Under Spinal Anesthesia — GSR electrodes will be connected before anaesthesia, and since the mother will be conscious during caesarean section, the newborn will have skin-to-skin contact with the mother immediately after birth. During this process, GSR signals of the mother and the baby will be recorded.
  Arms: Spinal Anestesia

SUMMARY:
A 2016 Cochrane Review shows that skin-to-skin contact promotes breastfeeding and strengthens mother-infant bonding. For the mother, skin-to-skin contact was found to promote early separation of the placenta, reduce postpartum haemorrhage, increase breastfeeding self-efficacy, reduce stress levels and promote oxytocin release. For the infant, it has been revealed that it provides important benefits such as decreased postnatal stress, improved thermoregulation, shortened crying time and increased breastfeeding success.

In line with this information, it is hypothesised that Galvanic Skin Response can be used to objectively evaluate the psychological and mental effects of early skin-to-skin contact on the mother and newborn after birth. The findings of this study will contribute to clinical practice by providing scientific evidence for neonatal care.

DETAILED DESCRIPTION:
This study will be carried out using galvanic skin response (GSR) to objectively evaluate the psychological and physiological effects of postnatal skin-to-skin contact on mother and infant. Scientific research shows that early postnatal skin-to-skin contact provides many benefits for both mother and baby. The 2016 Cochrane Review emphasises that skin-to-skin contact promotes breastfeeding and strengthens postnatal attachment. For the mother, skin-to-skin contact was found to promote early separation of the placenta, reduce postpartum haemorrhage, increase breastfeeding self-efficacy, support oxytocin release and reduce stress levels. In terms of the baby, it is seen that it has important benefits such as decreased postnatal stress, improved thermoregulation, shortened crying time and increased breastfeeding success. In the literature, the positive effects of skin-to-skin contact on the baby's body temperature, breastfeeding success and physiological stability have been proven.

This study will be conducted in Erciyes University Faculty of Medicine, Department of Obstetrics and Gynaecology and will be carried out with the participation of 100 volunteer mothers who will give birth by elective caesarean section at 37-40 weeks of gestation. In the study, two different groups, general anaesthesia and spinal anaesthesia, will be examined and the effects of anaesthesia type on skin-to-skin contact will be evaluated. After obtaining informed consent from the volunteer patients included in the study, their records will be created. Those who gave birth before 37 weeks of gestation, those who had normal vaginal delivery, those with known systemic diseases or fetal anomalies will be excluded from the study.

GSR electrodes will be connected to the mothers before anaesthesia and galvanic skin response will be measured during labour. After the baby is born, initial assessments will be made by the neonatal nurse and paediatrician and 1st and 5th minute APGAR scores will be determined. Cord pH value, birth weight and neonatal morbidity rates of the newborn will be recorded. The baby will be brought for skin-to-skin contact with the mother, and GSR signals from both mother and baby will be recorded during this process. Signal analyses will be performed by examining physiological changes during and after skin-to-skin contact with the newborn mother.

GSR signals will be recorded with the BIOPAC device. The measurements will be analysed by methods such as Short-Time Fourier Transform, Power Spectral Density and Wavelet Transform. Detailed analyses will be performed on the time-frequency axis using techniques such as Singular Spectrum Analysis and Empirical Mode Decomposition. In the classification phase, different algorithms such as artificial neural networks, support vector machines, logistic regression and clustering methods will be evaluated. FIR and IIR filtering methods will be applied in the processing of GSR signals to remove noise and interference from the signals.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy pregnancy between 37-40 weeks
2. Elective caesarean section
3. Having a singleton pregnancy

Exclusion Criteria:

1. Preterm labour under 37 weeks of gestation
2. Those with known systemic diseases
3. Those with known fetal anomalies
4. Pregnant women who will give birth normally
5. Multiple pregnancies

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Galvanic Skin Response | Effects of skin-to-skin contact with in 5 minutes after birth
  Skin To Skin contact of the newborn with the mother affects the Galvanic Skin Response.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Kayseri, Turkey (Türkiye)